CLINICAL TRIAL: NCT05091151
Title: Comparison of The Effectiveness of Intranasal Dexmedetomidine Sedation at Dose of 2 mcg/kg and 4 mcg/kg in Children Undergoing MRI at Cipto Mangunkusumo Hospital
Brief Title: Intranasal Dexmedetomidine Sedation at Dose of 2 mcg/kg Versus 4 mcg/kg in Children Undergoing MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Adhrie Sugiarto, dr. Adhrie Sugiarto, SpAn KIC, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes118
Record Dates: First submitted 2021-09-21; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia; Deep Sedation; Magnetic Resonance Imaging; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal dexmedetomidine at dose of 2 mcg/kg (Active Comparator): Subjects in IND 2 group received Intranasal dexmedetomidine at dose of 2 mcg/kg, before the MRI procedure through both nostrils using a 1 mL syringe. Patient was maintained in supine position for 1-2 minutes to maximize absorption.
  Interventions: Drug: Intranasal dexmedetomidine at dose of 2 mcg/kg and 4 mcg/kg
- Intranasal dexmedetomidine at dose of 4 mcg/kg. (Active Comparator): Subjects in IND 4 group received Intranasal dexmedetomidine at dose of 4 mcg/kg, before the MRI procedure through both nostrils using a 1 mL syringe. Patient was maintained in supine position for 1-2 minutes to maximize absorption.
  Interventions: Drug: Intranasal dexmedetomidine at dose of 2 mcg/kg and 4 mcg/kg

INTERVENTIONS:
Drug: Intranasal dexmedetomidine at dose of 2 mcg/kg and 4 mcg/kg — Intranasal dexmedetomidine were given 45 minutes before the MRI procedure through both nostrils using a 1 mL syringe.

SUMMARY:
This study aimed to compare the effectiveness of intranasal Dexmedetomidine sedation at Dose of 2 mcg/kg and 4 mcg/kg in Children Undergoing MRI at Cipto Mangunkusumo Hospital

DETAILED DESCRIPTION:
Ninety-four pediatric subjects who would undergo MRI with sedation were recruited. Subjects aged between 1-10 years old, ASA I-II, weighed between 1-30 kg were included in this study and assigned into two groups randomly. One group received 2 mcg/kg (IND2 group) and the other group received 4 mcg/kg (IND 4 group) of intranasal dexmedetomidine.

Randomization was done by the third party, who was not participated in the data collection, by using randomization tool from www.randomizer.org.

Dose of intranasal dexmedetomidine for each participant was concealed using closed envelope and was opened preprocedure by the second party who prepared the sedation drugs. The doctor, who gave sedation drug to the patient and recorded the data, was also blinded. All patients were blinded to data collection. Patients were allowed to drink clear fluid until 2 hours and required to fast for 6 hours before the procedure. Baseline heart rate, SpO2 was recorded premedication.

Subjects in IND 2 and IND 4 group received 2 mcg/kg and 4 mcg/kg intranasal dexmedetomidine. Intranasal drugs were given 45 minutes before the MRI procedure through both nostrils using a 1 mL syringe. Patient was maintained in supine position for 1-2 minutes to maximize absorption. After the patient was sedated, peripheral intravenous access was performed. The level of sedation was assessed using RSS. Heart rate, oxygen saturation, and RSS are recorded every 10 minutes until the procedure was done. After the target sedation has been reached, MRI started immediately. If the sedation target was not reached and/or the child moved, 0.5 mg/kg rescue dose of propofol would be given. After completing the MRI procedure, the patient was then transferred to the recovery room to record the recovery time. Outpatients were allowed to go home when they reached Aldrete score of 9-10.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 1-10 years old undergoing MRI
* ASA I-II
* Weighed between 1-30 kg

Exclusion Criteria:

* Patients who had history of hypersensitivity reaction to dexmedetomidine or showed an allergic reaction due to sedation drugs during MRI examination.
* Patients with cardiorespiratory, liver, kidney problems, risk of difficult airway, undergoing digoxin or beta blocker therapy, and failed to be sedated after 45 minutes since drug administered.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Onset sedation time of Intranasal dexmedetomidine. | 45 minutes before MRI procedure.
  This study compared the onset time of IND 2 to IND 4 group.
  Operational definition: Time taken from drug induction to achieve sedation (Ramsay sedation score 5).
  Ramsay Sedation Scoring system :
  1. Patient is anxious and agitated or restless, or both
  2. Patient is co-operative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response

SECONDARY OUTCOMES:
Duration of Sedation | During MRI procedure
  This study compared the duration of sedation of IND 2 to IND 4 group.
  Operational definition: Time taken from "achieving the sedation target" to "Ramsay's sedation score 3"
  Ramsay Sedation Scoring system :
  1. Patient is anxious and agitated or restless, or both
  2. Patient is co-operative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response

OTHER OUTCOMES:
Recovery time | Up to 2 hours after MRI procedure has been completed
  This study compared the recovery time in IND 2 to IND 4 group.
  Operational definition: Time calculated from the completion of the MRI procedure until the Aldrete score 9 is achieved
  (The Aldrete's scoring system is a commonly used scale for determining when patient can be safely discharged from the post-anesthesia care unit. A score of 8-10 is considered adequate to discharge a patient from Phase I of post anesthesia care.)
Adverse effect | During MRI procedure dan recovery time
  This study compared the adverse effect occured in IND 2 to IND 4 group.
  The acute side effects of sedation, including:
  Bradycardia (Heart Rate < 60 x/min and/or decrease in HR > 20% from baseline) Desaturation (Moderate desaturation if SpO2 < 95% for 15 seconds, Severe desaturation if SpO2 < 90% for 15 seconds) Allergic reaction (rash, itchy sensation, and hypotension)
Rescue dose of Propofol needed | During MRI procedure
  This study compared the amount of rescue dose of propofol needed in IND2 to IND4 group.
  This study calculated the amount of rescue dose of propofol needed during the MRI procedure under following conditions:
  If sedation targets are not achieved, inadequate, or the patient is immobile, boluses of propofol 0.5 mg/kg intravenously could be given to the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tug A, Hanci A, Turk HS, Aybey F, Isil CT, Sayin P, Oba S. Comparison of Two Different Intranasal Doses of Dexmedetomidine in Children for Magnetic Resonance Imaging Sedation. Paediatr Drugs. 2015 Dec;17(6):479-85. doi: 10.1007/s40272-015-0145-1. PMID 26323489
- [Result] Gupta A, Dalvi NP, Tendolkar BA. Comparison between intranasal dexmedetomidine and intranasal midazolam as premedication for brain magnetic resonance imaging in pediatric patients: A prospective randomized double blind trial. J Anaesthesiol Clin Pharmacol. 2017 Apr-Jun;33(2):236-240. doi: 10.4103/joacp.JOACP_204_16. PMID 28781452
- [Result] Olgun G, Ali MH. Use of Intranasal Dexmedetomidine as a Solo Sedative for MRI of Infants. Hosp Pediatr. 2018 Jan 23:hpeds.2017-0120. doi: 10.1542/hpeds.2017-0120. Online ahead of print. PMID 29363517
- [Result] Li BL, Zhang N, Huang JX, Qiu QQ, Tian H, Ni J, Song XR, Yuen VM, Irwin MG. A comparison of intranasal dexmedetomidine for sedation in children administered either by atomiser or by drops. Anaesthesia. 2016 May;71(5):522-8. doi: 10.1111/anae.13407. Epub 2016 Mar 3. PMID 26936022
- [Result] Schmitz A, Weiss M, Kellenberger C, O'Gorman Tuura R, Klaghofer R, Scheer I, Makki M, Sabandal C, Buehler PK. Sedation for magnetic resonance imaging using propofol with or without ketamine at induction in pediatrics-A prospective randomized double-blinded study. Paediatr Anaesth. 2018 Mar;28(3):264-274. doi: 10.1111/pan.13315. Epub 2018 Jan 27. PMID 29377404